CLINICAL TRIAL: NCT04692480
Title: A Pilot Study Assessing the Feasibility and Effectiveness of an Antepartum Breastfeeding Educational Video on In-Hospital and 6 Month Exclusive Breastfeeding Rates
Brief Title: A Pilot Study Assessing the Feasibility and Effectiveness of a Breastfeeding Educational Video on Breastfeeding Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Laurie Griffin, Obstetrics and Gynecology House Officer, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1539297
Record Dates: First submitted 2020-12-17; First posted 2020-12-31 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Breastfeeding, Exclusive
Keywords: Breastfeeding; Video education; Exclusive breastfeeding; Milk supply; Breastfeeding efficiency; Patient education; Antepartum
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Nulliparous women planning to exclusively breastfeed will be consented and will complete a survey regarding demographics and breastfeeding education experience. Participants will be randomized to viewing a standard breastfeeding education PDF (Control) or to watching an educational video entitled "Breastfeeding in the First Hour, It's in Your Hands"(Intervention group). Both activities will occur on a tablet. Participants will undergo routine intrapartum care. On the day of discharge, patient's will complete a survey that includes the Breastfeeding Self-Efficiency Scale-Short Form, the Perception of Insufficient Milk Questionnaire, and questions regarding in hospital breastfeeding educational experiences. Data will be compared between the two groups to determine if antepartum video education improved perception of breast milk supply and efficiency and increases exclusive breastfeeding rates. At 6 months postpartum, women will be surveyed by phone regarding their breastfeeding status.
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding Video Education (Experimental): Participants will view a breastfeeding educational video entitled "Breastfeeding in the First Hour, It's in Your Hands."
  Interventions: Behavioral: Breastfeeding Video Education
- Control (Other): Participants will view a PDF of breastfeeding education materials available for inclusion in standard discharge paper work.
  Interventions: Behavioral: Breastfeeding PDF education

INTERVENTIONS:
Behavioral: Breastfeeding Video Education — Video entitled "Breastfeeding in the First Hour, It's in Your Hands"
  Arms: Breastfeeding Video Education
Behavioral: Breastfeeding PDF education — PDF of standard breastfeeding education handouts
  Arms: Control

SUMMARY:
Given the known health benefits of breast milk, the World Health Organization and pediatric and obstetrical professional societies all recommend that babies only consume breast milk (also referred to as "exclusive breastfeeding (EBF)") through 6 months of age. While many women initiate breastfeeding while at the study institution hospital, the rate of exclusive breastfeeding when mothers and babies are discharged is only 34%. Sixty percent of mothers stopped breastfeeding earlier than intended to primarily due to concerns about difficulty with lactation (i.e. sore nipples, inadequate milk supply), baby's nutrition (i.e weight gain and satiety) and effort required to pump breast milk. It is known that prenatal education by trained health care providers is effective in increasing EBF rates; however, these interventions are time and labor intensive and require employment of breastfeeding specialists. Therefore, a simple, brief, easily accessible breastfeeding education tool is needed to directly educated new mothers on how to breastfeed and what the actual nutritional needs of an infant are in order to support women's breastfeeding goals. The objective of this study is to assess whether a simple breastfeeding education video viewed at the time of admission to the hospital for delivery will increase EBF at the time of hospital discharge through 6 months postpartum by improving women's perception of their milk supply and their breast feeding efficiency.

The investigators predict that woman who view a short breastfeeding education video just prior to delivery will have an improved perception of their breastfeeding efficiency and milk supply and will be more likely to avoid formula use while admitted to the hospital and though 6 months postpartum. In this study, the investigators will randomly assign women to view an educational video focused on breastfeeding in the first days of a baby's life and compare them to women who receive the standard educational pamphlet on breastfeeding given to all women delivering at the study institution. The investigators will then survey each participant after her delivery on how she is feeding her baby (breast milk, formula, or both) and how she perceives her milk supply and breastfeeding efficiency just before she is discharged from the hospital. The investigators will then call women on the phone at 6 weeks, 3 months and 6 months to reassess how they are feeding their babies (breast milk, formula or both). In addition to baseline characteristics about the individuals such as age, race, and employment status, information regarding their pregnancy and delivery will be obtained to assess for any confounding factors that may effect their ability to breastfeed. This research will help determine if video education can provide sufficient education to help increase breastfeeding rates. Additionally, this research may inform the research community on the overall effectiveness of video education in healthcare, allowing for a similar approach to be used for other educational initiatives.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous woman
* >18 years of age
* Fluency in English or Spanish
* Intention to exclusively breastfeed
* Admitted to Women and Infants Hospital (Providence, RI) for induction of labor, labor, or primary cesarean delivery.
* Gestational age between 37'0-42'0

Exclusion Criteria:

* Prior breastfeeding experience (ex: induced lactation for prior child)
* Contraindications to breastfeeding,
* Intention to utilize formula
* Extremis prohibiting consent
* Women who require Intensive Care Unit (ICU) admission, whose infants require Neonatal Intensive Care Unit (NICU) admission, or who suffer an intrapartum fetal demise or neonatal death will be excluded from final analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Breastfeeding rates at hospital discharge | 1-4 days Postpartum
  Using a self reported survey of infant feeding practices including exclusive breastfeeding, breastfeeding with formula supplementation or formula feeding only, the investigators aim to determine if participants who viewed the breastfeeding education video had increased breastfeeding rates compared to women who viewed the control PDF materials at time of hospital discharge.
Maternal perception of breastfeeding efficiency at hospital discharge | 1-4 days Postpartum
  Using the validated Breastfeeding Self-Efficiency Scale-Short Form, a Likert scale survey ranging from 1 (not confident at all) to 5 (very confident), the investigators aim to determine if maternal perception of breastfeeding efficiency at time of hospital discharge is increased for women who viewed the breastfeeding video compared to those who viewed the control PDF materials.
Maternal perception of milk supply at hospital discharge | 1-4 days Postpartum
  Using the validated Perception of Insufficient Milk Questionnaire, a Likert scale survey ranging from 1 (strongly disagree) to 10 (strongly agree) the investigators aim to determine if maternal perception of milk supply at time of hospital discharge is increased for women who viewed the breastfeeding video compared to those who viewed the control PDF materials. Outcome will be measured on the Likert scale.

SECONDARY OUTCOMES:
Breastfeeding rates at 6 weeks postpartum | 6 weeks postpartum
  Using a self reported phone survey of infant feeding practices including exclusive breastfeeding, inclusively breastfeeding with formula supplementation, formula feeding only, or solid food supplementation, the investigators aim to determine if participants who viewed the breastfeeding education video had increased breastfeeding rates compared to women who viewed the control PDF materials at 6 weeks postpartum.
Breastfeeding rates at 3 months postpartum | 3 months postpartum
  Using a self reported phone survey of infant feeding practices including exclusive breastfeeding, inclusively breastfeeding with formula supplementation, formula feeding only, or solid food supplementation, the investigators aim to determine if participants who viewed the breastfeeding education video had increased breastfeeding rates compared to women who viewed the control PDF materials at 3 months postpartum.
Breastfeeding rates at 6 months postpartum | 6 months postpartum
  Using a self reported phone survey of infant feeding practices including exclusive breastfeeding, inclusively breastfeeding with formula supplementation, formula feeding only, or solid food supplementation, the investigators aim to determine if participants who viewed the breastfeeding education video had increased breastfeeding rates compared to women who viewed the control PDF materials at 6 months postpartum.
Maternal perceptions of acceptability of breastfeeding education interventions | 1-4 days Postpartum
  To determine if women find breastfeeding educational interventions during delivery hospitalization to be acceptable and helpful Using a self reported survey of women's experience with breastfeeding support resources during hospital admission, the investigators aim to determine if the video or control education was acceptable and helpful to participants. Outcome will be measured on the Likert scale from 1 (not helpful at all) to 5 (very helpful).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie B Griffin, MD/PhD, Principal Investigator — Women and Infants Hospital/Brown Univerisity
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, we do not plan to make IPD available.

REFERENCES:
- See also: Breastfeeding educational Video "Breastfeeding in the First Hour, It's in Your Hands" in English — https://firstdroplets.com/downloads
- See also: Breastfeeding educational Video "Breastfeeding in the First Hour, It's in Your Hands" in Spanish — https://es.firstdroplets.com/descargas/